CLINICAL TRIAL: NCT04251936
Title: Modification of Alternative Reward Cue Reactivity and Cognitive Control Through Physical Activity in Human Tobacco Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Ströhle, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRR265 C03
Record Dates: First submitted 2020-01-16; First posted 2020-02-05 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Healthy; Tobacco Use Disorder
Keywords: tobacco use disorder; fMRI; physical exercise; reward system; cognitive control
MeSH Terms: conditions — Tobacco Use Disorder; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training plus smoking cessation group program (Experimental)
  Interventions: Behavioral: Exercise training; Behavioral: Smoking cessation group program
- Smoking cessation group program (Active Comparator)
  Interventions: Behavioral: Smoking cessation group program

INTERVENTIONS:
Behavioral: Exercise training — The moderate-intense aerobic exercise training will involve supervised aerobicycle ergometer training for 30 min with 60-80% HRmax three times per week for 12 weeks.
  Arms: Exercise training plus smoking cessation group program
Behavioral: Smoking cessation group program — Participants of both groups will receive a 6-week standard cognitive behavioral therapy-oriented smoking cessation group program (SCP, one 60 min session per week).

SUMMARY:
This study investigates the mechanisms, through which physical exercise impacts positively on abstinence in tobacco use disorder, with fMRI and behavioral tests.

DETAILED DESCRIPTION:
This study will test the hypothesis that physical exercise training modifies alternative reward cue reactivity and cognitive control in tobacco use disorder and that these modifications mediate the effect of exercise on abstinence. Continued physical exercise training was shown to reduce tobacco consumption and prevent relapse in tobacco use disorder (TUD). However, the psychological and neural mechanisms through which exercise training exerts its effects on tobacco consumption are not clear. The aim of this project is to identify the effects of a 12-week aerobic exercise training in TUD and to test how these exercise-related changes may mediate the effect of exercise training on abstinence. Investigations will focus on two potential mechanisms of regaining control: (1) modifications of tobacco and alternative reward cue reactivity and (2) improvement of cognitive control. Two aspects of cognitive control will be addressed: inhibitory control and cognitive down-regulation of craving. It is expected, first, that exercise training (compared to standard treatment) leads to desensitization towards tobacco cues and sensitization towards alternative reward cues, reflected in altered craving and neural (fMRI) cue reactivity. Second, it is expected that exercise training will lead to increased cognitive control (i.e., inhibitory control and cognitive down-regulation of craving), reflected in increased activation of prefrontal control regions (fMRI). Third, it is expected that effects of exercise on abstinence will be mediated by sensitization towards alternative reward cues and enhanced cognitive control. In an exploratory manner, gender differences in the effects of exercise training will be studied. Understanding the psychological and neural underpinnings will help to optimize and individualize exercise trainings in TUD.

ELIGIBILITY:
Inclusion Criteria:

* Tobacco use disorder according to DSM-5
* right-handedness
* sufficient ability to communicate with investigators
* ability to provide informed consent and to use self-rating scales
* seeking treatment for TUD
* no contra-indication for aerobic exercise

Exclusion Criteria:

* severe internal or neurological comorbidities
* axis I mental disorders other than TUD (except for mild depression, adjustment disorder and specific phobias) in the last 12 months according to DSM-5
* history of brain injury
* pregnancy
* exclusion criteria for MRI
* positive drug screening (opioids, benzodiazepines, cocaine, amphetamines)
* psychotropic medication within the last 14 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in nicotine consumption from pre-intervention to post-intervention | Pre-intervention and post-intervention (up to 2 weeks after intervention end)
  self-report
Change in nicotine consumption from pre-intervention to follow-up | Pre-intervention and follow-up (12 weeks after intervention end)
  self-report
Change in BOLD during cue reactivity task (fMRI) from pre-intervention to post-intervention | Pre-intervention and post-intervention (up to 2 weeks after intervention end)
  Blood Oxygen Level Dependent especially within the ventral striatum, the ventral medial prefrontal cortex and the amygdala during a cue reactivity task with neutral, tobacco, alternative reward images and warning images depicting aversive consequences of smoking
Change in BOLD during down-regulation of craving task (fMRI) from pre-intervention to post-intervention | Pre-intervention and post-intervention (up to 2 weeks after intervention end)
  Blood Oxygen Level Dependent especially within the ventral striatum, the amygdala and the dorsolateral prefrontal cortex during a cognitive down-regulation of craving task with tobacco and alternative reward stimuli
Change in BOLD during stop-signal task (fMRI) from pre-intervention to post-intervention | Pre-intervention and post-intervention (up to 2 weeks after intervention end)
  Blood Oxygen Level Dependent especially within the dorsolateral prefrontal cortex during a stop signal task
Change in craving ratings (behavioral) from pre-intervention to post-intervention | Pre-intervention and post-intervention (up to 2 weeks after intervention end)
  The participants' answers to the question "how strong is your desire to consume the item shown" on a scale of 1 - 8 is averaged over a total of 144 pictures of nicotine and alternative reward stimuli. The change in average ratings between pre-intervention and post-intervention is computed.
Change in down-regulation of craving (behavioral) from pre-intervention to post-intervention | Pre-intervention and post-intervention (up to 2 weeks after intervention end)
  The down-regulation of craving task is carried out as described in Kober et al., 2010. As described there, the down-regulation of craving is calculated as the difference in craving ratings between the now and later condition (20 nicotine and alternative reward stimuli are shown in the now and later condition). The change in the down-regulation of craving between pre- and post-intervention is then calculated.
Change in stop-signal reaction time (behavioral) from pre-intervention to post-intervention | Pre-intervention and post-intervention (up to 2 weeks after intervention end)
  Stop-signal reaction time in the stop-signal task

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Background] Kober H, Mende-Siedlecki P, Kross EF, Weber J, Mischel W, Hart CL, Ochsner KN. Prefrontal-striatal pathway underlies cognitive regulation of craving. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14811-6. doi: 10.1073/pnas.1007779107. Epub 2010 Aug 2. PMID 20679212
- [Derived] Kunas SL, Stuke H, Plank IS, Laing EM, Bermpohl F, Strohle A. Neurofunctional alterations of cognitive down-regulation of craving in quitting motivated smokers. Psychol Addict Behav. 2022 Dec;36(8):1012-1022. doi: 10.1037/adb0000820. Epub 2022 Feb 17. PMID 35175067